CLINICAL TRIAL: NCT03877315
Title: Patient Reported Outcome After Stemmed Versus Stemless Total Shoulder Arthroplasty for Glenohumeral Osteoarthritis: a Patient Blinded Randomized Clinical Trial
Brief Title: Patient Reported Outcome After Stemmed Versus Stemless Total Shoulder Arthroplasty for Glenohumeral Osteoarthritis.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Zealand University Hospital (Other)
Collaborators: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Zaid Issa, Medical doctor, shoulder and elbow surgeon., Zealand University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REG-106-2018
Record Dates: First submitted 2019-03-12; First posted 2019-03-15 (Actual); Last update posted 2022-12-22 (Actual); Status verified 2022-12

CONDITIONS: Shoulder Pain; Shoulder Osteoarthritis; Shoulder Arthritis
MeSH Terms: conditions — Shoulder Pain

STUDY DESIGN:
Who Masked: Participant
Masking Description: Patients will be blinded to which implant type they are receive. This will be done by not sharing the operation chart files with the patient's online file records; the inserted shoulder prosthesis will be noted by a unique code in operation file, and the radiologist will be asked not to describe the post-operation x-ray controls.
  The primary investigator will conduct the blinded statistical analysis supervised by the biostatistician.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Stemmed (Active Comparator): Subjects operated with stemmed shoulder arthroplasty, Biomet Comprehensive® Total Shoulder System.
  Interventions: Device: Stemmed shoulder arthroplasty, Biomet Comprehensive® Total Shoulder System.
- Non-Stemmed (Active Comparator): Subjects operated with stemless shoulder arthroplasty, Biomet Comprehensive® Nano Shoulder System.
  Interventions: Device: Stemless shoulder arthroplasty, Biomet Comprehensive® Nano Shoulder System.

INTERVENTIONS:
Device: Stemmed shoulder arthroplasty, Biomet Comprehensive® Total Shoulder System. — A total shoulder prosthesis used in treating glenohumeral osteoarthritis
  Arms: Stemmed
Device: Stemless shoulder arthroplasty, Biomet Comprehensive® Nano Shoulder System. — A total shoulder prosthesis used in treating glenohumeral osteoarthritis
  Arms: Non-Stemmed

SUMMARY:
Stemless shoulder arthroplasty systems with uncemented metaphyseal fixation have been used in Europe for glenohumeral osteoarthritis since 2004. The stemless design has several theoretical advantages compared with the stemmed shoulder arthroplasty systems: restoring patients' anatomy, preserving humeral bone stock, and few complications in component removal if the need for a revision arthroplasty arises. The purpose of the study is to compare the short-term, patient-reported outcome of stemless and stemmed total shoulder arthroplasty.

DETAILED DESCRIPTION:
Glenohumeral joint osteoarthritis is a common cause of shoulder pain, affecting up to one-third of patients older than 60 years. Surgical treatment is indicated for patients with glenohumeral arthritis who continue to experience significant symptoms despite an appropriate course of non-operative management. Shoulder arthroplasty accounts for the third most common joint replacement procedure after the hip and knee arthroplasty. Based on data from the National Patient Registry, The Statistical Department of the Danish National Board of Health, the use of primary shoulder replacement in Denmark increased from 12 replacements per 100,000 inhabitants in 2005 to 19 replacements per 100,000 inhabitants in 2015. Glenohumeral osteoarthritis is now the most common indication for shoulder arthroplasty in Denmark.

Many different shoulder arthroplasty designs are available on the market. The stemless shoulder arthroplasty system with uncemented metaphyseal fixation has been used in Europe for glenohumeral osteoarthritis since 2004. The indications for anatomical stemless TSA are the same as for anatomical stemmed TSA: osteoarthritis, rheumatoid arthritis, and post-traumatic osteoarthritis or osteonecrosis.

The contraindications for anatomical stemless TSA are acute proximal humerus fracture, inadequate metaphyseal bone stock, and rotator cuff insufficiency.

Stemless TSA has several theoretical advantages over stemmed TSA: restoring patients' anatomy (humeral shaft angle, humeral head diameter, and lateralization); preserving humeral bone stock, and few complications in component removal should the need of a revision arthroplasty arise. A recent review of 3,360 anatomical total shoulder arthroplasties found an overall complication rate of 10.3%. Periprosthetic fractures accounted for 6.7% and humeral component loosening for 1.4% of all complications. Complications related to the stemmed humeral component can be divided into intraoperative (malpositioning, false route, periprosthetic fracture) and postoperative (loosening, migration, disassembly, periprosthetic fracture, stem fracture) complications. When a revision is necessary because of infection or periprosthetic fracture, the removal of a well-fixed or cemented humeral component can be challenging and lead to bone damage.

Few outcome studies on stemless TSA are available. A recent review of 11 observational studies (published 2010-2016), incorporating a total of 929 patients, reported comparable short- and midterm functional outcomes between stemmed and stemless shoulder prosthesis. Otherwise, there are few well-conducted and adequately powered clinical studies.

The objective of this study is to increase knowledge about shoulder function after operation with anatomical TSA by comparing the patient-reported outcome after stemmed and stemless anatomical TSA for glenohumeral osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged ≥ 18 years.
2. Patients have been referred to the Orthopedic Department or Zealand University Hospital, Koege or Hvidovre University Hospital for shoulder pain during the study period.
3. Patients have the ability to read trial information in Danish and give informed consent.
4. The diagnosis will be based on plain radiographs (at least two perpendicular views), reduction of joint space, and/or osteophyte formation.
5. Clinical presentation with pain at night and/or daily pain, pain in overhead activity, and consumption of pain medication.

Exclusion Criteria:

1. Previous shoulder surgery that involves the humeral head and/or the glenoid cavity.
2. Patients with alcohol or drug abuse problems that can compromise rehabilitation and follow-up appointments as assessed by the recruiting surgeon at the first visit.
3. Patients unable to understand instructions in Danish, follow the rehabilitation protocol, or answer the questionnaires because of physical or cognitive inabilities as evaluated by the recruiting surgeon at the first visit.
4. Brachial plexus palsy.
5. Patients with previous fractures around the shoulder (clavicle, scapula, and proximal humerus fractures).
6. Patients with MRI scan-verified full thickness total tear of one or more of the rotator cuff tendons.
7. Patients with CT scan-verified glenoid retroversion ≥ 20° that does not allow glenoid component fixation without bone graft or need an augmented glenoid component.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
Western Ontario Osteoarthritis of the Shoulder Score (WOOS) | 12 months after surgery
  The WOOS is a patient-administered, disease-specific ques¬tionnaire for measurement of the quality of life of patients with osteoarthritis. It provides scores for four domains: (1) physical symptoms; (2) sport, recreation, and work; (3) lifestyle; and (4) emotions. Patients answer each question using the visual analogue scale. The WOOS score is calculated by measuring the distance from the left side of the line and calculating the possible score ranging from 0 to 100 (recorded to the nearest 0.5 mm.) It consists of 19 questions, and the total score ranges from 0 to 1900. A maximum score of 1900 signifies that the patient has an extreme decrease in shoulder-related quality of life, whereas a score of 0 signifies that the patient has no decrease in shoulder-related quality of life. The questionnaire has been translated into Danish and validated and tested on patients with shoulder osteoarthritis.

SECONDARY OUTCOMES:
Western Ontario Osteoarthritis of the Shoulder Score (WOOS) | 3 months after surgery
Oxford Shoulder Score (OSS) | 3 and 12 months after surgery
  Oxford Shoulder Score (OSS) is a measurement tool for the assessment of outcomes of shoulder surgery. It has been tested and validated in patients with primary or secondary osteoarthritis. The OSS is a 12-item questionnaire, with each item scored from 0-4; thus, the overall score is the sum of the scores received for individual questions. This results in a continuous score ranging from 0 (most severe symptoms) to 48 (least severe symptoms). For simplicity of presentation, the raw scores will be converted to a percentage of the maximum score. We will use a validated Danish version.
EQ-5D questionnaire | 3 and 12 months after surgery
  The EQ-5D, the health status component of the EuroQol assessment (EuroQol Group, Rotterdam, The Netherlands), is a generic instrument for describing and evaluating health-related quality of life. The EuroQol instrument has been designed for self-completion by the respondent.
  The EQ-5D is a descriptive system comprising five dimensions in each of which the respondents describe their health state: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has five levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. The patient choose one of five levels for each dimension, and thus a five-digit number (EuroQol Group 1990) can define the resulting health state. We received permission to use the Danish version (permission ID number 27296).

CONTACTS AND LOCATIONS:
Overall Officials: Zaid Issa, MD, Principal Investigator — Zealand University Hospital Koege
Locations (1):
- Zealand University Hospital, Køge, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Issa Z, Rasmussen JV, Petersen JK, Schantz K, Brorson S. Patient-reported outcome after stemmed versus stemless total shoulder arthroplasty for glenohumeral osteoarthritis: a patient-blinded randomized clinical trial. Trials. 2019 Jul 12;20(1):427. doi: 10.1186/s13063-019-3535-9. PMID 31300025